CLINICAL TRIAL: NCT04480762
Title: A Randomised, Double Blind, Placebo Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-1703 Injection Administered Subcutaneously in Healthy Subjects
Brief Title: A Trial of SHR-1703 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1703-101
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SHR-1703-Subcutaneous administration of Dose 1 (Experimental): A single subcutaneous injection of SHR-1703 (Dose 1) or Placebo
  Interventions: Drug: SHR-1703; Drug: Placebo
- SHR-1703-Subcutaneous administration of Dose 2 (Experimental): A single subcutaneous injection of SHR-1703 (Dose 2) or Placebo
  Interventions: Drug: SHR-1703; Drug: Placebo
- SHR-1703-Subcutaneous administration of Dose 3 (Experimental): A single subcutaneous injection of SHR-1703 (Dose 3) or Placebo
  Interventions: Drug: SHR-1703; Drug: Placebo
- SHR-1703-Subcutaneous administration of Dose 4 (Experimental): A single subcutaneous injection of SHR-1703 (Dose 4) or Placebo
  Interventions: Drug: SHR-1703; Drug: Placebo
- SHR-1703-Subcutaneous administration of Dose 5 (Experimental): A single subcutaneous injection of SHR-1703 (Dose 5) or Placebo
  Interventions: Drug: SHR-1703; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1703 — SHR-1703
Drug: Placebo — Placebo of the SHR-1703

SUMMARY:
SHR-1703 is a monoclonal antibody under development for severe asthma. This study is the first study in Healthy subjects. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of a single dose SHR-1703 administered subcutaneously in Chinese healthy subjects.

DETAILED DESCRIPTION:
This study will be conducted at 1 study center in China. Approximately 42 healthy Chinese male and female subjects, aged 18 to 55 inclusive, will be randomized to receive a single SC administration of SHR-1703: Treatment 1, Treatment 2, Treatment 3, Treatment 4 and Treatment 5. Each subject will participate in only 1 treatment group. The total length of the study for each subject is up to 190 days (28 days of screening and 155+/- 7 days of further study visits).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Able to read, comprehend and write at a sufficient level to complete study materials.
* Aged 18 to 55 years (inclusive).
* Body weight equal or more than 45.0 kg and BMI within the range between 19 and 24kg/m2 (inclusive).
* AST, ALT, alkaline phosphatase and bilirubin equal or less than ULN.
* Healthy Chinese as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the Jiangsu HengRui Medicine Co Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subjects must commit to consistent and correct use of an acceptable method of birth control from the start of trial to the next month after the last visit.
* A negative pre-study drug/alcohol screen.

Exclusion Criteria:

* Allergy/intolerance to the SHR-1703 and/or excipients in the formulation, or any other Biologics
* Positive Hepatitis B surface antigen or positive Hepatitis C antibody or human immunodeficiency virus - HIV antibody or Syphilis serological test at screening
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to screening in the current study: 3 months, 5 half-lives or fellow-up period of the investigational product (whichever is longer).
* Use of any medicines, including prescription or Over-the-Counter drugs (including herbal and dietary supplements, not including regular vitamins and paracetamol which be used occasionally in the recommended dose) within 1 month or 5 half-lives (whichever is longer) prior to the administration.
* Subjects who have received immune inhibitors within 6 months prior to screening
* Subjects who have had severe trauma or surgery within 6 months prior to screening, or who plan to undergo surgery during the trial.
* Blood donation history within 1 month prior to screening ,or severe blood loss(total blood volume≥400 ml)，or blood transfusion within 2 months
* Subjects who are inoculated live (attenuated) vaccine within 1 month prior to screening or during the trial.
* Subject who is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* At the discretion of the investigator, a subject will not be eligible for this study if he/she is in the following cases: the subject is not able to complete the study, or present a significant risk to the subject, or present other factors(e.g. infirmity. etc.) that may prevent the enrolment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse events (AEs) and serious adverse events (SAEs) | From Day 1 to Days 155
  The number and percentage of subjects with treatment-emergent AE/SAE/AE by severity/drug-related AE/drug-related SAE/death in each dose level group and overall. AE/SAE will be displayed by MedDRA SOC and/or PT
Safety as determined by abnormality in haematology | From Day 1 to Days 155
  Measurement of red blood cell count, white blood cell count, haemoglobin and platelets
Safety as determined by abnormality in clinical chemistry | From Day 1 to Days 155
  Measurement of kidney function (e.g.urea ,creatinine, Uric acid), liver function(ALP, ALT, AST, albumin, total bilirubin), lipid profile(total cholesterol, triglycerides), ions.
Safety as determined by abnormality in urinalysis | From Day 1 to Days 155
  Measurement of glucose, ketones, leukocytes, blood and protein
Safety as determined by evaluation of blood pressure in mmHg | From Day 1 to Days 155
  Measurement of blood pressure (systolic and diastolic in mmHg)
Safety as determined by evaluation of Pulse rate in beats per minute | From Day 1 to Days 155
  Measurement of Pulse rate in beats per minute
Safety as determined by evaluation of body temperature in degree Celsius | From Day 1 to Days 155
  Measurement of body temperature in degree Celsius
Safety as determined by evaluation of Respiratory rate in beats per minute | From Day 1 to Days 155
  Measurement of Respiratory rate in beats per minute
Safety as determined by analysis of 12-lead ECG variables: heart rate (beats per minute) | From Day 1 to Days 155
  The ECG variables will be summarized by absolute value at each visit by treatment group, together with the corresponding changes from baseline.
Safety as determined by analysis of 12-lead ECG variables: PR, QRS, QT and QTcF (milliseconds) | From Day 1 to Days 155
  The ECG variables will be summarized by absolute value at each visit by treatment group.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | From Day 1 to Follow-UP ( Days2, Days 3,Days 4, Days 5, Days 6, Days 8, Days 11, Days 15, Days 22 , Days 29, Days 43, Days 64, Days 92, Days 120, Days 155)
  To assess the Pharmacokinetic profile of Subcutaneously administration of SHR-1703 in healthy Chinese subjects.
Time to maximum observed concentration (tmax) | From Day 1 to Follow-UP ( Days2, Days 3,Days 4, Days 5, Days 6, Days 8, Days 11, Days 15, Days 22 , Days 29, Days 43, Days 64, Days 92, Days 120, Days 155)
  To assess the Pharmacokinetic profile of Subcutaneously administration of SHR-1703 in healthy Chinese subjects.
Area under the concentration-time curve from 0 to the last measurable time point (AUC0-t) | From Day 1 to Follow-UP ( Days2, Days 3,Days 4, Days 5, Days 6, Days 8, Days 11, Days 15, Days 22 , Days 29, Days 43, Days 64, Days 92, Days 120, Days 155)
  To assess the Pharmacokinetic profile of Subcutaneously administration of SHR-1703 in healthy Chinese subjects.
Area under the concentration-time curve from 0 to infinity (AUC0-∞) | From Day 1 to Follow-UP ( Days2, Days 3,Days 4, Days 5, Days 6, Days 8, Days 11, Days 15, Days 22 , Days 29, Days 43, Days 64, Days 92, Days 120, Days 155)
  To assess the Pharmacokinetic profile of Subcutaneously administration of SHR-1703 in healthy Chinese subjects.
Apparent clearance (CL/F) | From Day 1 to Follow-UP ( Days2, Days 3,Days 4, Days 5, Days 6, Days 8, Days 11, Days 15, Days 22 , Days 29, Days 43, Days 64, Days 92, Days 120, Days 155)
  To assess the Pharmacokinetic profile of Subcutaneously administration of SHR-1703 in healthy Chinese subjects.
Apparent volume of distribution at terminal phase (Vz/F) | From Day 1 to Follow-UP ( Days2, Days 3,Days 4, Days 5, Days 6, Days 8, Days 11, Days 15, Days 22 , Days 29, Days 43, Days 64, Days 92, Days 120, Days 155)
  To assess the Pharmacokinetic profile of Subcutaneously administration of SHR-1703 in healthy Chinese subjects.
Time for concentration to decrease by 50% (concentration half-life) (t1/2) | From Day 1 to Follow-UP ( Days2, Days 3,Days 4, Days 5, Days 6, Days 8, Days 11, Days 15, Days 22 , Days 29, Days 43, Days 64, Days 92, Days 120, Days 155)
  To assess the Pharmacokinetic profile of Subcutaneously administration of SHR-1703 in healthy Chinese subjects.
Anti-drug antibody (ADA) as determined by evaluation of ADA positive percentage and ADA negative percentage | From Day 1 to Follow-UP ( Days 8, Days 15, Days 29, Days 92, Days 120, Days 155)
  To assess the immunogenicity of SHR-1703

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang L, Fang Y, Luo Y, Fu M, Shen K, Luo Z. Safety, pharmacokinetics and pharmacodynamics of SHR-1703, an innovative long-acting anti-interleukin-5 monoclonal antibody, in healthy subjects: a randomized, double-blind, dose-escalation, placebo-controlled phase I study. Expert Opin Investig Drugs. 2024 Jul;33(7):741-752. doi: 10.1080/13543784.2024.2361065. Epub 2024 Jun 3. PMID 38805242